CLINICAL TRIAL: NCT06189391
Title: An Open-Label, Dose Escalation Phase 1a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of MK-1045 (CN201) in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate MK-1045 (CN201) in Participants With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma (MK-1045-001/CN201-101)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MSD R&D (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1045-001; MK-1045-001 (Other: MSD); CN201-101 (Other: Curon Biopharmaceutical Co., LTD)
Record Dates: First submitted 2023-08-30; First posted 2024-01-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MK-1045 Fixed Dose (Experimental): Participants will receive MK-1045 via intravenous (IV) infusion on Day 1 of each week for 3 consecutive weeks followed by one week off of each four-week cycle for up to 12 months until discontinuation or death.
  Interventions: Drug: MK-1045
- MK-1045 Step-up Dose (Experimental): Participants will receive MK-1045 via an IV infusion in a step-up dose with priming once a week (Q1W) for a 3-week cycle for up to 12 months until discontinuation or death.
  Interventions: Drug: MK-1045

INTERVENTIONS:
Drug: MK-1045 — IV infusion
  Other Names: CN201

SUMMARY:
Researchers are looking for new ways to treat people with relapsed or refractory B-Cell Non-Hodgkin Lymphoma (B-NHL). B-cells are a type of white blood cells that make antibodies and help fight infections. Non-Hodgkin Lymphoma is a type of cancer in the lymphatic system causing enlarged lymph nodes and/or organs in belly or chest. Relapsed means a disease or condition comes back after treatment Refractory means a disease does not respond to treatment or stops responding to a treatment.

MK-1045, the study medicine, is designed to treat relapsed or refractory B-NHL. MK-1045 is an immunotherapy, which is a treatment that helps the immune system fight cancer.

This is the first study in which MK-1045 will be given to people. The goal of this study is to learn about:

* The safety of MK-1045 and how well people tolerate it.
* The highest dose of MK-1045 that is well tolerated.
* How well MK-1045 works to treat relapsed or refractory B-NHL.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Inclusion Criteria

Inclusion Criteria include, but are not limited to:

* Has relapsed or refractory B-cell Non-Hodgkin's lymphoma (B-NHL) with disease history meeting the following World Health Organization (WHO) diagnostic subtypes of B-NHL that are CD19-positive in pathologic Immunohistochemistry test: diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL) (Grade I to III), marginal zone lymphoma, lymphoplasmacytic lymphoma, mantle cell lymphoma, small lymphocytic lymphoma, and transformed large B-cell lymphoma (During the dose-escalation phase, participants other than those treated with Chimeric antigen receptor T-cell (CAR-T) who cannot provide proof of pathologic immunohistochemistry CD19 positivity but have previous proof of CD20 positivity may be considered for enrollment after discussion with the sponsor)

  * Relapse is defined as the occurrence of progressive disease (PD) after complete response (CR) or partial response (PR) has been achieved after adequate treatment. Note: For DLBCL participants, relapse must occur after participants undergoing at least two lines of therapy; for other participants, they must undergo at least one line of therapy.
  * Refractory is defined as a situation that there is no standard of care available or that it is not applicable to use standard of care at this stage, including: Participants who are unresponsive to standard of care (e.g., monotherapy or combination therapy containing anti-CD20 monoclonal antibody) and whose best response to standard therapy is PD or stable disease (SD); Participants who are not eligible for autologous hematopoietic stem cell transplantation (ASCT) and have relapsed PD after receiving ASCT; Participants who have failed on chimeric antigen receptor T cell (CAR-T) immunotherapy, but the first dose of the study intervention must be at least 3 months after discontinuation of CAR-T therapy, and CD19 positive expression is still present in tumor tissue.
* Has at least one evaluable tumor lesion per the Lugano 2014 criteria, i.e., a lymph node lesion > 15 mm in long diameter or an extranodal lesion > 10 mm in long diameter according to computed tomography (CT) cross-sectional imaging or magnetic resonance imaging (MRI)
* Has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2 and an estimated survival time of more than 3 months
* Has essentially normal: bone marrow function; coagulation function; liver function; kidney function; lung function; and heart function

Exclusion Criteria

Exclusion Criteria include, but are not limited to:

* Has any other non-Hodgkin lymphoma (NHL) not listed in inclusion criteria
* Has been treated with anti-CD3/CD19 bispecific antibody (BsAb) prior to first dose of study intervention
* Has received chemotherapy, endocrine therapy, radiotherapy (palliative radiotherapy 2 weeks prior to the first administration of the investigational drug), or biologic therapy, and small molecule targeted agents within 2 weeks prior to the first administration of the investigational drug or within 5 half-lives of the drug, whichever is shorter
* Has received anti-CD20 antibody or anti-CD19 antibody within 4 weeks prior to first use of the investigational drug
* Has received anti-tumor immunotherapy or other unlisted clinical study intervention within 4 weeks prior to the first dose of study intervention, or within 5 half-lives of the drug, whichever is shorter
* Has undergone any major organ surgery (excluding aspiration biopsy) or significant trauma within 4 weeks prior to the first dose of study intervention or those requiring elective surgeries during the study
* Has received systemic corticosteroids (prednisone >10 mg/day or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of the study intervention, excluding the following agents: topical, ocular, intra-articular, intranasal, and inhaled corticosteroids, and short-term, prophylactic use of corticosteroids (e.g. to prevent radio contrast agent induced allergic reactions)
* Has used immunomodulatory agents, including but not limited to thymosin, interleukin-2 (IL-2), interferon (IFN) and anti-tumor Chinese patent drugs or Chinese herbal medicines within 14 days prior to the first dose of study intervention
* Has had a live attenuated vaccines within 4 weeks prior to the first dose of study intervention
* Has a central nervous system (CNS) infiltration
* Has previous or concomitant CNS diseases, including epilepsy, hemorrhagic/ischemic stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disorder, organic cerebellar syndrome, or mental diseases
* Has prior or concomitant malignancies (except cured basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, prostatic intraepithelial neoplasia, and other tumors that have been clinically cured for 5 years as assessed by the investigator)
* Has uncontrolled active infections currently requiring systemic anti-infective therapy within 3 days prior to first dose
* Has active hepatitis B and/or hepatitis C. Participants who are positive for antibodies to hepatitis C virus (HCV). Participants who are hepatitis B surface antigen (HBsAg) positive are not allowed to enroll in the dose-escalation period; however, those who were hepatitis B surface antigen (HBsAg)-positive but hepatitis B Virus deoxyribonucleic acid (HBV DNA)-negative and adherent to entecavir antiviral therapy and who agreed to regular monthly monitoring of HBV DNA are allowed to enroll in the dose-expansion period
* Has a history of immunodeficiency, including testing positive for human immunodeficiency virus (HIV) antibody
* Has a history of serious cardiovascular and cerebrovascular disease, including but not limited to: severe cardiac rhythm or conduction abnormalities; acute coronary syndrome, congestive heart failure, stroke, or other Grade 3 or higher cardiovascular and cerebrovascular events within 6 months prior to the first dose; ≥ Class II cardiac function as per New York Heart Association (NYHA) functional class or LVEF < 50%; or clinically uncontrollable hypertension
* Has previous or current interstitial lung disease
* Has acute graft-versus-host disease (GVHD) or active chronic GVHD at present
* Has active or history of autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis, etc.) that may relapse, or participants who are at risks (e.g., organ transplant requiring immunosuppressive therapy). Participants with the following diseases are allowed to be further screened for enrollment: hypothyroidism managed with hormone replacement therapy only, and skin diseases not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia).
* Has received immunotherapy with known Grade 3 or higher immune-related adverse events (irAEs)
* Has non-hematologic adverse reactions from prior anti-tumor therapy have not recovered to Grade ≤ 1 as assessed by National Cancer Institute NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 (excluding toxicities such as alopecia that are assessed by the investigator to have no safety risk)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience a Dose-limiting Toxicity (DLT) | Up to ~28 Days
  DLT are any of the following drug related (DR) investigator-assessed adverse events: Grade 4 neutropenia that does not recover to Grade ≤ 2 after more than 5 days of supportive care including granulocyte colony-stimulating factor (G-CSF), or ≥ Grade 3 febrile neutropenia; Grade 4 platelet (PLT) decreased, or Grade 3 PLT decreased with bleeding; Grade 4 anemia. Grade 4 non-hematologic toxicity; Grade 3 non-hematologic toxicity that does not recover to Grade ≤ 2 within 3 days after best supportive care (excluding simple laboratory abnormalities without clinical significance as assessed by the investigator). Participants with ≥ Grade 3 tumor lysis syndrome who recover to ≤ Grade 2 within 14 days after optimal supportive therapy will be excluded from the definition of DLT. A DLT was also any other toxic reactions requiring permanent discontinuation of the study intervention.
Number of Participants who Experience an Adverse Event (AE) | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. The number of participants who experience an AE will be reported.
Number of Participants who Experience a Serious Adverse Events (SAE) | Up to ~15 months
  An SAE refers to an untoward medical occurrence such as death, life-threatening event, permanent or serious disability or loss of function, need for hospitalization or prolongation of hospitalization after the participant receives the intervention, and congenital abnormalities or birth defects. The number of participants who experience a SAE will be reported.
Number of Participants who Experience a Drug-related Adverse Event (DRAE) | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. A DRAE is defined as an AE definitely related, probably related, or possibly related to the study intervention. The number of participants who have experienced a DRAE will be reported.
Number of Participants who Experience an AE of Grade 3 or higher | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the study intervention, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. AEs are graded on a scale from 1-5 with 1=Mild, 2=Moderate, 3=Severe or medically significant but not immediately life-threatening, 4= Life threatening consequences, and 5=Death due to AE. The number of participants who experience an AE of grade 3 or above will be presented.
Number of Participants who Experience an AE for Each Severity Grade from 1-5 | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the study intervention, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. AEs are graded on a scale from 1-5 with 1=Mild, 2=Moderate, 3=Severe or medically significant but not immediately life-threatening, 4= Life threatening consequences, and 5=Death due to AE. The number of participants who experience an AE in each category of AEs from 1-5 will be presented.
Number of Participants who Experience a SAE or Serious Drug-related AE | Up to ~15 months
  An SAE refers to an untoward medical occurrence such as death, life-threatening event, permanent or serious disability or loss of function, need for hospitalization or prolongation of hospitalization after the participant receives the study intervention, and congenital abnormalities or birth defects. A drug related SAE is defined as an SAE definitely related, probably related, or possibly related to the study intervention. The number of participants who experience a SAE or a serious drug-related AE will be reported.
Number of Participants who Experience a Dose Modification Due to an AE or DRAE | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the study intervention, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. A drug related AE includes AEs definitely related, probably related, and possibly related to the study intervention. The number of participants who experience a dose modification due to an AE or DRAE will be presented.
Number of Participants who Withdraw from the Study due to an AE or DRAE | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the study intervention, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. A drug related AE includes AEs definitely related, probably related, and possibly related to the study intervention. The number of participants who discontinue the study due to an AE will be presented.
Number of Participants who Died due to an AE or DRAE | Up to ~15 months
  An AE is defined as any untoward medical event that occurs after a participant receives the study intervention, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the study intervention. A drug related AE includes AEs definitely related, probably related, and possibly related to the study intervention. The number of participants who died due to an AE or DRAE will be presented.

SECONDARY OUTCOMES:
Mean Change in Serum MK-1045 Concentration After Administration | Baseline and up to 12 months
  Blood samples will be collected to determine the mean change from baseline in serum concentration of MK-1045.
Area Under the Concentration-time Curve (AUC) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the AUC of MK-1045 in plasma.
Area Under the Concentration-time Curve from Time 0 to 168 Hours Post Dose (AUC0-168) of MK-1045 | Pre-dose and at designated time points post-dose up to 168 hours
  Blood samples will be collected to determine the AUC0-168 of MK-1045 in plasma.
Area Under the Concentration-time Curve from Time 0 to Last Quantifiable Concentration Post Dose (AUC0-last) of MK-1045 | Pre-dose and at designated time points post-dose up to 168 hours
  Blood samples will be collected to determine the AUC0-last of MK-1045 in plasma.
Maximum Concentration (Cmax) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the Cmax of MK-1045 in plasma.
Time to Maximum Concentration (Tmax) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the Tmax of MK-1045 in plasma.
Terminal Elimination Half-life (T1/2) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the t1/2 of MK-1045 in plasma.
Clearance (CL) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the CL of MK-1045 in plasma.
Concentration at the End of Dosing Interval (Ctrough) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the Ctrough of MK-1045 in plasma.
Area Under the Concentration-time Curve from Time 0 to the Dosing Interval (168 Hours) at Steady State (AUC0-tau) of MK-1045 | Pre-dose and at designated time points post-dose up to 168 hours
  Blood samples will be collected to determine the AUC0-tau of MK-1045 in plasma.
Accumulatio Ratio Based on Cmax (RAC-Cmax) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the RAC_Cmax of MK-1045 in plasma.
Accumulation Ratio Based on AUC0-tau (RAC_AUC0-tau) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the RAC-AUC0-tau of MK-1045 in plasma.
Steady State Clearance (CLss) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the CLss of MK-1045 in plasma.
Steady State Apparent Volume of Distribution (Vss) of MK-1045 | Pre-dose and at designated time points post-dose up to 12 months
  Blood samples will be collected to determine the Vss of MK-1045.
Mean Number of B Cells in Peripheral Blood After Administration of MK-1045 | Baseline and up to 12 months
  Blood samples will be collected to determine the mean number of B cells in peripheral blood after treatment with MK-1045.
Mean Number of T cells in Peripheral Blood After Administration of MK-1045 | Baseline and up to 12 months
  Blood samples will be collected to determine the mean number of T cells in peripheral blood after treatment with MK-1045.
Mean Level of T Cell Activation After Administration with MK-1045 | Baseline and up to 12 months
  Blood samples will be collected to determine the mean T cell activation after treatment with MK-1045.
Mean Level of T Cell Proliferation After Administration of MK-1045 | Baseline and up to 12 months
  Blood samples will be collected to determine the mean level of T cell proliferation after treatment with MK-1045.
Mean Level of Cytokines in Peripheral Blood After Administration of MK-1045 | Baseline up to 12 months
  Blood samples will be collected to determine the mean level of cytokines after treatment with MK-1045.
Percentage of Participants who Develop Anti-drug Antibodies (ADA) to MK-1045 | Baseline and up to 15 months
  Blood samples will be collected to determine the percentage of participants with ADAs to MK-1045 after treatment with MK-1045.
Objective Response Rate (ORR) | Up to 15 months
  ORR is defined as the percentage of the participants who had complete response (CR) or partial response (PR) and will be evaluated using computed tomography (CT) and positron emission tomography (PET)-CT. Response will be assessed based on the International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). The percentage of participants who experience CR or PR will be presented.
Duration of Response (DOR) | Up to ~15 months
  For participants who demonstrate a CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. Participants will be evaluated using CT and metabolic imaging (FDG-PET). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). DOR will be presented among participants who demonstrated CR or PR.
Complete Response Rate (CRR) | Up to ~15 months
  CRR is defined as the percentage of the participants who had complete response (CR) and will be evaluated using computed tomography (CT) and positron emission tomography (PET)-CT. Response will be assessed based on the International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. The percentage of participants who experience a CR will be presented.
Duration of Complete Response (DCR) | Up to ~15 months
  For participants who demonstrate a CR, DCR is defined as the time from the first documented evidence of CR until disease progression or death due to any cause, whichever occurs first. Participants will be evaluated using CT and metabolic imaging (FDG-PET). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. DCR for participants with CR will be presented.
Progression Free Survival (PFS) | Up to ~15 months
  PFS is defined as the time from first dose to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PD per Lugano criteria is defined as new or increased adenopathy, splenic volume increase, new or larger non-measured lesions, recurrent previously resolved lesions, new extranodal lesion >1 cm in any axis, a new node >1.5 cm in any axis. PFS will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (15):
- China (15):
  - Fifth Medical Center of PLA General Hospital ( Site 0005), Beijing, Beijing Municipality
  - Beijing Cancer hospital ( Site 0001), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 0011), Xiameng, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 0003), Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University. ( Site 0004), Shijiazhuang, Hebei
  - Henan Cancer Hospital ( Site 0009), Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University ( Site 0006), Zhengzhou, Henan
  - Jiangxi Cancer Hospital ( Site 0007), Nanchang, Jiangxi
  - The First Hospital Of Jilin University ( Site 0014), Changchun, Jilin
  - Shandong Cancer Hospital ( Site 0008), Jinan, Shandong
  - Fudan University Shanghai Cancer Center ( Site 0012), Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University ( Site 0013), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 0002), Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital. ( Site 0018), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 0010), Tianjinc, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com